CLINICAL TRIAL: NCT02556567
Title: Exploring the Effects of Sleep Patterns and Physical Activity on Asthma in Adolescents With Wrist-worn Smart Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: University of Arkansas (Other); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 204310
Record Dates: First submitted 2015-09-08; First posted 2015-09-22 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Asthma
Keywords: Sleep patterns; Physical activity; Fitbit
MeSH Terms: conditions — Asthma; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Other): Participants will wear the Fitbit® Charge Heart Rate (HR) wristband for eight weeks.
  Interventions: Other: Fitbit® Charge Heart Rate (HR) wristband

INTERVENTIONS:
Other: Fitbit® Charge Heart Rate (HR) wristband — The Investigators will conduct a proof of concept and feasibility study to explore associations between asthma symptoms and sleep patterns and physical activity over an 8-week intervention period among 20 adolescent patients with persistent asthma.

SUMMARY:
This is a research study to find associations between asthma symptoms and sleep patterns and physical activity among adolescent patients with persistent asthma. The Investigators will collect Fitbit® sensor data and survey data from each adolescent enrolled in the study.

DETAILED DESCRIPTION:
Investigators from the University of Arkansas for Medical Sciences (Pediatrics), the University of Arkansas at Little Rock and the University of Florida will work together to conduct a research study to find associations between asthma symptoms, sleep patterns, and physical activity over an 8-week period among adolescent patients with persistent asthma.

The goal of this research study is to find new ways for teenagers to manage their asthma. Full understanding of the connection and interference of sleep patterns and physical activity with asthma symptoms will be very helpful for teenagers with asthma to better manage their daily routine and asthma care. This research study will use wrist-worn devices (i.e. Fitbit® wristbands) to collect participants' sleep and physical activity data.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 14 and ≤ 17 years;
2. Teen access to a mobile smartphone device with a data plan or a computer with reliable internet connection, compatible with the Fitbit® application during the study period;
3. Diagnosis of mild, moderate or severe persistent asthma per National Heart Lung Blood Institute (NHLBI).

Exclusion Criteria:

1. Current smokers and adolescents with significant underlying respiratory disease other than asthma (such as cystic fibrosis) that could potentially interfere with asthma-related outcome measures;
2. Prior diagnosis of sleep disorder;
3. Patients with significant co-morbid conditions (such as moderate to severe developmental delay) that could interfere with the adolescent's ability to self-monitor asthma;
4. Inability to speak or understand English (child or parent).

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Asthma Symptoms , Sleep Patterns and Physical Activity | 8 weeks
  Fitbit built-in sensors (e.g., accelerometer, gyroscope, and heart rate sensors will measure disruptive sleep patterns, decreased levels of physical activity and asthma symptoms using response pattern scoring from baseline for 8 weeks.

SECONDARY OUTCOMES:
Risk of Increasing Asthma Symptoms | 8 weeks
  Identify risks of increasing asthma symptoms based on daily Fitbit® data from baseline over an 8 week time period.

OTHER OUTCOMES:
Machine Learning Techniques | 8 weeks
  Develop techniques to explore associations between Fitbit® data and patient reported outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara T. Perry, MD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data. We will disseminate our research findings in medical sponsored journals, presentations and posters.

REFERENCES:
- [Result] Moorman JE, Rudd RA, Johnson CA, King M, Minor P, Bailey C, Scalia MR, Akinbami LJ; Centers for Disease Control and Prevention (CDC). National surveillance for asthma--United States, 1980-2004. MMWR Surveill Summ. 2007 Oct 19;56(8):1-54. PMID 17947969
- [Result] Akinbami LJ, Moorman JE, Garbe PL, Sondik EJ. Status of childhood asthma in the United States, 1980-2007. Pediatrics. 2009 Mar;123 Suppl 3:S131-45. doi: 10.1542/peds.2008-2233C. PMID 19221156
- [Result] Calmes D, Leake BD, Carlisle DM. Adverse asthma outcomes among children hospitalized with asthma in California. Pediatrics. 1998 May;101(5):845-50. doi: 10.1542/peds.101.5.845. PMID 9565412
- [Result] Smaldone A, Honig JC, Byrne MW. Sleepless in America: inadequate sleep and relationships to health and well-being of our nation's children. Pediatrics. 2007 Feb;119 Suppl 1:S29-37. doi: 10.1542/peds.2006-2089F. PMID 17272582
- [Result] Walker TJ, Reznik M. In-school asthma management and physical activity: children's perspectives. J Asthma. 2014 Oct;51(8):808-13. doi: 10.3109/02770903.2014.920875. Epub 2014 May 14. PMID 24796650
- [Result] Meltzer LJ, Ullrich M, Szefler SJ. Sleep duration, sleep hygiene, and insomnia in adolescents with asthma. J Allergy Clin Immunol Pract. 2014 Sep-Oct;2(5):562-9. doi: 10.1016/j.jaip.2014.02.005. Epub 2014 Apr 13. PMID 25213049
- [Result] Wanrooij VH, Willeboordse M, Dompeling E, van de Kant KD. Exercise training in children with asthma: a systematic review. Br J Sports Med. 2014 Jul;48(13):1024-31. doi: 10.1136/bjsports-2012-091347. Epub 2013 Mar 23. PMID 23525551